CLINICAL TRIAL: NCT04275323
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety and Efficacy of NL003 in Subject With Critical Limb Ischemia(Rutherford 4)
Brief Title: Safety and Efficacy Study Using Gene Therapy for Critical Limb Ischemia (NL003-CLI-III-1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Northland Biotech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL003-CLI-III-1
Record Dates: First submitted 2020-01-18; First posted 2020-02-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-03

CONDITIONS: Arterial Occlusive Disease; Ischemia; Ulcers; Peripheral Vascular Disease
Keywords: HGF; Gene; Critical Limb Ischemia
MeSH Terms: conditions — Arterial Occlusive Diseases; Ischemia; Ulcer; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- investigational produc (Experimental): Patients in this treatment group will receive 8mg NL003 respective in D0、14、28
  Interventions: Genetic: NL003
- Placebo (Placebo Comparator): Patients in this group will receive normal saline respective in D0、14、18
  Interventions: Other: Normal Saline

INTERVENTIONS:
Genetic: NL003 — Day 0: 8mg of NL003 (32 injections of 0.5ml of NL003) Day 14: 8mg of NL003 (32 injections of 0.5ml of NL003) Day 28: 8mg of NL003 (32 injections of 0.5ml of NL003)
  Other Names: HGF plasmid; pCK-HGF-X7
  Arms: investigational produc
Other: Normal Saline — Day 0: 16ml of Normal Saline (32 injections ) Day 14: 16ml of Normal Saline (32 injections ) Day 28: 16ml of Normal Saline (32 injections )
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of recombinant human hepatocyte growth factor (HGF) bare plasmid injection for local intramuscular injection in the treatment of patients with severe lower limb hemorrhagic disease (Rutherford grade 4)

DETAILED DESCRIPTION:
Management of CLI process consumes a significant amount of healthcare resources,and the new therapeutic approaches are required.

Hepatocyte growth factor (HGF) has been shown to be a potent angiogenic growth factor stimulating the growth of endothelial cells and migration of vascular smooth muscle cells. Because of its pluripotent capabilities, increasing the availability of HGF in ischemic tissues to achieve therapeutic angiogenesis has been a growing area of research.

This study will use NL003, which is a DNA plasmid that contains novel genomic cDNA hybrid human HGF coding sequence (HGF-X7) expressing two isoforms of HGF, HGF 728 and HGF 723. As there are currently no approved drugs that can reverse CLI and as most patients have exhausted surgical and endovascular intervention options, inducing angiogenesis in the affected limb with NL003 may result in an increase in tissue perfusion, which, in turn improve wound healing, reduce pain and improve limb salvage rates.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 20 and 80 (when signing informed consent), both male and female;

  2. Patients diagnosed with lower limb arterial ischemic disease based on DSA or CTA and combined with their medical history and clinical manifestations and Rutherford grade 4 (resting pain) must meet the following criteria simultaneously (if both limbs of the subject have lower limb arterial ischemic disease, the researcher shall choose one limb for the study).Resting ankle systolic pressure (dorsal foot artery or posterior tibial artery) ≤70mmHg or ABI≤0.5 or TcPO2 < 30mmHg;In the first 3 months after randomized inclusion, DSA or CTA confirmed severe stenosis (≥70%) or occlusion of superficial femoral artery or popliteal artery or inferior knee artery.

  3. Chronic lower limb arterial ischemia combined with resting pain met the following requirements: resting pain lasted for more than 2 weeks when the informed consent was signed;

  4. Agreed to use the basic treatment drugs as required during the trial, and recorded the daily record of the subjects in a timely and complete manner. The compliance of the basic treatment drugs and the subjects' diary filling during the screening period was 70%.

  5. Agree to use appropriate contraceptive measures during the experiment;Female subjects of reproductive age, blood pregnancy test negative;

  6. Signed informed consent

Exclusion Criteria:

* 1. Patients with acute lower limb ischemia or acute exacerbation of chronic lower limb ischemia.

  2. Vascular reconstruction (bypass or intravascular therapy) or sympathetic resection or amputation was performed within 4 weeks prior to the signing of the informed consent.

  3. Due to surgical operation, the patient is still in the postoperative risk period, and the researcher judges that the patient is not suitable for the test.

  4. Main-iliac artery stenosis 70%.

  5. Patients with ischemic ulcer of lower extremity.

  6. NYHA classification of cardiac function is classified as grade (see annex 1 for specific classification criteria).

  7. Patients with unstable angina pectoris due to cerebral infarction, cerebral hemorrhage and myocardial infarction within 3 months before signing the informed consent.

  8. Refractory hypertension (taking three or more antihypertensive drugs, systolic blood pressure 180mmHg or diastolic blood pressure 110mmHg).

  9. Proliferative retinopathy and retinopathy examination is not available.

  10. Inability to accurately describe symptoms and emotions.

  11. Severe liver disease with uncompensated cirrhosis, jaundice, ascites or hemorrhagic varices.

  12. Current recipients of immunosuppressants or chemoradiotherapy.

  13. Anti-hiv antibody positive, anti-hepatitis c antibody positive and hepatitis b surface antigen positive (if the subject is HBsAg positive and HBV DNA in peripheral blood is combined, the researcher believes that the subject's chronic hepatitis b is stable and will not increase the risk of the subject, the subject can be selected).

  14. Results of laboratory examination during screening period: hemoglobin <80g/L, white blood cell count < 3.0109 /L, platelet <75 109/L, upper limit of normal AST or ALT> 3 times, upper limit of normal serum creatinine > 2.5 times, or other laboratory examination indicators appear abnormal that researchers think may affect the evaluation of test results.

  15. Patients with poor blood glucose control after treatment (hemoglobin a1c >10%).

  16. Previously diagnosed with malignant tumor, or any of the following test results determined by the investigator to be at risk of tumor: fecal occult blood test;Chest X-ray examination or chest CT examination;Alpha-fetoprotein (AFP), carcinoembryonic antigen (CEA) and ca19-9;Male subjects, prostate specific antigen test (PSA, free PSA);Female subjects, cervical smear (Pap), mammography/b-ultrasound and ca-125 examination;The investigators determined that additional tests were necessary to eliminate the tumor risk.

  17. In the opinion of the investigators, patients with comorbidities that affect safety and efficacy evaluation, or with a predicted survival of less than 12 months.

  18. Frequent drinkers within the 12 months prior to the signing of the informed consent, i.e., those who drank more than 14 units of alcohol per week (1 unit =360 mL beer or 45 mL alcohol of 40% spirits or 150 mL wine) or substance abusers.

  19. Participate in other clinical trials within 3 months before signing the informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Complete pain relief rate | Day180
  1.Day180 visit (5-7 days prior to visit, including the visit day), mean daily pain score was 0；2.A pain score of 0 must be measured without the use of analgesics.

SECONDARY OUTCOMES:
The time when the pain completely goes away | Day180
  The time when the pain completely goes away.
Complete pain relief rate | Day90
  Day90 visit (5-7 days prior to visit, including the visit day), mean daily pain score was 0.
Changes in site visits, pain scores after use of the study drug | Day14,Day28,Day60,Day90,Day120,Day180
  The Numerical Rating Scale（NRS） was used to record changes in pain in subjects, who chose a number that best represented their pain in the past 24 hours, ranging from 0 (painless) to 10 (the most intense pain imaginable).The NRS scale is pain free (0), mild pain (1-3), moderate pain (4-6), and severe pain (7-10).
Percent of Participants with a 50% reduction in pain score from baseline | Day180
  Percent of Participants with a 50% reduction in pain score from baseline.
The type and dose of analgesics varied from baseline | Day14,Day28,Day60,Day90,Day120,Day180
  The types and dosages of analgesics varied from baseline at each site after the use of the study drug.
Changes in Rutherford grading from baseline to Day180 | Day14,Day28,Day60,Day90,Day120,Day180
  The severity of critical Limb ischemia was assessed by Rutherford grading at screening, D14, D28, D60, D90, and D180, respectively.Rutherford grades chronic limb ischemic disease into grades 0 to 6, of which 4, 5 and 6 are chronic severe ischemia.
Changes in quality of life scores from baseline to Day180 | Day14,Day28,Day60,Day90,Day120,Day180
  The WHOQOL-BREF was conducted to evaluate the subjective perception of Critical Limb Ischemia, including the subjects' perception of quality of life, health, or other aspects of life.The whoqol-bref has 26 questions. Each question is rated on a scale of 1 to 5, with 1 for poor quality of life and 5 for good quality of life.
Changes in the ABI from the baseline to Day180 | Day60,Day90,Day120,Day180
  Ankle-brachial index (ABI) refers to the ratio of systolic blood pressure of the anterior tibial artery (dorsal foot artery) or posterior tibial artery to the systolic blood pressure of the brachial artery.Participants were tested for ankle-brachial index (ABI).The normal value of ABI is 0.9-1.4, where <0.4 is severe ischemia,0.41-0.9 is mild to moderate ischemia, and ABI>1.4 indicates vascular wall calcification.
Percentage of patients who underwent revascularization (open surgery or interventional therapy) had a large amputation rate and mortality | Day180
  Day180, percentage of patients undergoing revascularization (open surgery or interventional therapy) major amputation rate mortality.

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Beijing Hospitai, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Ninth People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xuzhou Mining Group General Hospital, Xuzhou, Jiangsu
  - Chifeng Municipal Hospital, Chifeng, Neimenggu
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai seventh people's hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - First Affiliated Hospital of Xi 'an Jiaotong University, XiAn, Shanxi
  - Second Affiliated Hospital of Xi 'an Jiaotong University, XiAn, Shanxi